CLINICAL TRIAL: NCT02646124
Title: Adding Diazepam to Standard Management of Acute, Non-radicular Low Back Pain. An Emergency Department Based Randomized Comparative Effectiveness Study
Brief Title: Diazepam Use With Standard Management for Acute Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, principal investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-4639
Record Dates: First submitted 2015-12-31; First posted 2016-01-05 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Low Back Pain
Keywords: benzodiazepine
MeSH Terms: conditions — Low Back Pain | interventions — Naproxen; Diazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Diazepam (Experimental): Naproxen +Diazepam
  Interventions: Drug: Naproxen; Drug: Diazepam
- Placebo (Active Comparator): Naproxen + Placebo
  Interventions: Drug: Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Naproxen 500mg by mouth two times a day, #20
Drug: Placebo — 28 placebo capsules
  Other Names: Placebo Diazepam
  Arms: Placebo
Drug: Diazepam — Diazepam 5mg capsules, 1-2 tabs by mouth two times a day, #28
  Arms: Diazepam

SUMMARY:
Given the poor pain and functional outcomes that persist beyond an Emergency Department (ED) visit for musculoskeletal low back pain (LBP), we propose a clinical trial to evaluate whether combining a benzodiazepine with an NSAID is more effective than nonsteroidal antiinflammatory drug (NSAID) monotherapy for the treatment of acute, non-traumatic, non-radicular low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) causes 2.4% of visits to US emergency departments (ED) resulting in 2.7 million visits annually. In general, outcomes for these patients are poor. One week after ED discharge, 70% of patients report persistent back-pain related functional impairment and 69% report analgesic use within the previous 24 hours. Three months after the ED visit, 48% of these patients report functional impairment, 42% report moderate or severe pain, and 46% report persistent analgesic use.

It is not clear how acute LBP should be treated. Non-steroidal anti-inflammatory drugs (NSAID) are guideline-supported, first line therapy for acute LBP. NSAIDs are more efficacious than placebo with regard to pain relief, global improvement, and requirement of analgesic medication but are not sufficient therapy for as many as ½ of ED patients, who continue to suffer despite therapy with NSAIDs. Treatment of LBP with multiple concurrent medications is common in the ED--emergency physicians often prescribe benzodiazepines, skeletal muscle relaxants, or opioids in combination with NSAIDs. However, work recently completed here at Montefiore has revealed that combining skeletal muscle relaxants or opioids with NSAIDs does not improve outcomes. It remains uncertain if adding benzodiazepines to NSAIDs improves LBP outcomes.

Although benzodiazepines are used in 300,000 US ED visits for LBP annually, scant evidence exists to determine the appropriateness of this approach. Efficacy of benzodiazepines may be related to direct or centrally-mediated action on skeletal muscle or may instead work by mitigating anxiety about the condition or numbing a patient to the pain.

Given the poor pain and functional outcomes that persist beyond an ED visit for musculoskeletal LBP, we propose a clinical trial to evaluate whether combining a benzodiazepine with an NSAID is more effective than NSAID monotherapy for the treatment of acute, non-traumatic, non-radicular low back pain. Specifically, we will evaluate the following hypothesis:

A daily regimen of naproxen + diazepam will provide greater relief of LBP than naproxen + placebo one week after an ED visit, as measured by the Roland Morris Disability Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Present to ED primary for management of LBP, defined as pain originating between the lower border of the scapulae and the upper gluteal folds. Flank pain, that is pain originating from tissues lateral to the paraspinal muscles, will not be included.
* Absence of non-musculoskeletal etiology of low back, such as urinary tract infection, cystic ovarian disease, or influenza like illness. The primary clinical diagnosis, at the conclusion of the ED visit, must be a diagnosis consistent with non-traumatic, non-radicular, musculoskeletal LBP.
* Patient is to be discharged home. Patients admitted to the hospital are more likely to be treated with parenteral medication and therefore are not appropriate for this study.
* Age 21-69 Enrollment will be limited to adults younger than 70 years because of the increased risk of adverse medication effects in the elderly.
* Non-radicular pain: pain cannot radiate below the gluteal folds in a radicular pattern. Patients with non-radicular pain extending below the gluteal folds will not be excluded
* Pain duration <2 weeks (336 hours). Patients with more than two weeks of pain are at increased risk of poor pain and functional outcomes.(2)
* Prior to the acute attack of LBP, back pain cannot have occurred once per month or more frequently. Patients with more frequent back pain are at increased risk of poor pain and functional outcomes.(2)
* Non-traumatic LBP: no substantial and direct trauma to the back within the previous month
* Functionally impairing back pain: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* -Not available for follow-up
* Pregnant or breast-feeding
* Chronic pain syndrome defined as use of any analgesic medication on a daily or near-daily basis
* Allergic to or intolerant of investigational medications
* Contra-indications to non-steroidal anti-inflammatory drugs: peptic ulcer disease, history of gastro-intestinal bleeding, congestive heart failure, advanced renal disease, aspirin sensitive asthma
* Contra-indications to diazepam: glaucoma, myasthenia gravis, cirrhosis, sleep apnea, history of alcoholism or substance abuse

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diazepam | Placebo
Started | 57 | 57
Completed | 57 | 55
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Diazepam: Naproxen +Diazepam
  Naproxen: Naproxen 500mg by mouth two times a day, #20
  Diazepam: Diazepam 5mg capsules, 1-2 tabs by mouth two times a day,, #28
- Total: Total of all reporting groups
Arm/Group | Diazepam | Placebo | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34 (12) | 38 (12) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 30 | 33 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 57 | 114
Duration of Back Pain Prior to Study [Median (Inter-Quartile Range); unit: hours] | 72 [24 to 108] | 48 [12 to 96] | 48 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment as Measured by the Roland Morris Disability Questionnaire
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life. The change in RMDQ is obtained by subtracting the RMDQ score at one week after discharge from the baseline score.
Time Frame: Between baseline and one week after emergency department discharge
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 57 | 55
units on a scale | 11 [9 to 13] | 11 [9 to 13]

2. Secondary Outcome: Number of Participants With Moderate or Severe Pain, as Measured on an Ordinal Scale
Description: Patients with moderate or serve pain. Worst Lower Back Pain (LBP) over the previous 24 hours, using a four point ordinal scale: severe, moderate, mild, or none.
Time Frame: 1 week after discharge from emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 57 | 55
Participants | 18 | 12

3. Secondary Outcome: Number of Participants Who Required Analgesic Medication for Low Back Pain Within the Previous 24 Hours
Description: Telephone questionnaire is used to assess patients needing any analgesic or low back pain medication within the previous 24 hours.
Time Frame: One week after discharge from the emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 57 | 55
Participants | 26 | 25

4. Secondary Outcome: Number of Participants Who Required Analgesic Medication for Low Back Pain Within the Previous 72 Hours
Description: Patients needing any analgesic or LBP medication within the previous 72 hours
Time Frame: Assessed three months after emergency department discharge
Population: data not collected
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Participants Satisfied With Treatment
Description: Participants who answered "Yes" when asked the question "Do you want to receive the same combination of medications during a subsequent visit to the ER?"
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 57 | 55
Participants | 44 | 37

ADVERSE EVENTS:
Arm/Group | Diazepam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/55
Other Adverse Events (participants affected / at risk) | 12/57 | 8/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diazepam (N=57) | Placebo (N=55)
Drowsy (Nervous system disorders) | 4 (4) | 1 (1)
Dizzy (Nervous system disorders) | 1 (1) | 0 (0)
Stomach irritation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Other (General disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes